CLINICAL TRIAL: NCT00441545
Title: A Prospective, Multicenter, Open-label, Randomized, Cross-over Study to Compare the Efficacy and Safety of Fosrenol® and Sevelamer Hydrochloride in Patients Receiving Hemodialysis for End Stage Renal Disease
Brief Title: Head to Head Study Against Sevelamer Hydrochloride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-319; 2006-004959-38 (EudraCT Number)
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Disease, Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — lanthanum carbonate; Sevelamer

ARMS (2):
- 1 (Experimental): Fosrenol (Lanthanum carbonate)
  Interventions: Drug: Fosrenol (Lanthanum Carbonate)
- 2 (Active Comparator): Sevelamer hydrochloride
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: Fosrenol (Lanthanum Carbonate) — The starting dose is a total daily dose of 2250mg of Fosrenol (Lanthanum carbonate) to a maximum dose of 3000mg daily. Chewable tablets will be administered orally with meals in 750mg and 1000mg strength tablets.
  Other Names: FOSRENOL
  Arms: 1
Drug: Sevelamer hydrochloride — The starting dose is a total daily dose of 4800mg of sevelamer hydrochloride up to a maximum of 6400 mg daily. Sevelamer hydrochloride 800mg tablets, administered orally with meals.
  Arms: 2

SUMMARY:
To compare the efficacy of Fosrenol (Lanthanum carbonate) and sevelamer hydrochloride in the reduction of serum phosphorus levels from baseline.

DETAILED DESCRIPTION:
To compare the efficacy of Fosrenol (Lanthanum carbonate) and sevelamer hydrochloride in the reduction of serum phosphorus levels from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Adults with end stage renal disease who are receiving dialysis

Exclusion Criteria:

* Subjects with significant gastrointestinal disorders
* Subjects who are pregnant or nursing
* Subjects currently taking lanthanum carbonate, sevelamer hydrochloride, cinacalcet hydrochloride
* Subjects who are HIV positive
* Subjects with clinical significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-01-05 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (44):
- United States (34):
  - DSI Renal Inc., Mesa, Arizona
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - Southwest Kidney Institute, PLC, Tempe, Arizona
  - Tempe, Arizona
  - University of Arizona Health Service Center, Tucson, Arizona
  - Clinical Research Connections, Jonesboro, Arkansas
  - South Valley Dialysis Center, Encino, California
  - VA Greater Los Angeles Health Care System, West LA, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - North Valley Nephrology, Yuba City, California
  - Western Nephrology & Metabolic Bone Disease, PC, Thornton, Colorado
  - Shands University of Florida Outpatient Dialysis, Gainesville, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Pines Clinical Research, Pembroke Pines, Florida
  - Clinical Research Center of Indian River Medical Center, Vero Beach, Florida
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Renal Physicians of Georgia, Macon, Georgia
  - Evanston Northwestern Hospital, Evanston, Illinois
  - Research by Design, LLC, Evergreen Park, Illinois
  - Nephrology Inc., Mishawaka, Indiana
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Creighton University Medical Center, Omaha, Nebraska
  - Hypertension and Nephrology, Associates, Eatontown, New Jersey
  - Winthrop Dialysis Center, Mineola, New York
  - SUNY at Stony Brook NY, Stony Brook, New York
  - Wake Nephrology Associates, Raleigh, North Carolina
  - Southeastern Nephrology Associates, Wilmington, North Carolina
  - Northwest Renal Clinic, Portland, Oregon
  - Carolina Nephrology, PA, Greenville, South Carolina
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
  - Rosa Verde Tower, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio Medicine/Nephrology, San Antonio, Texas
  - Alexandria Kidney, Alexandria, Virginia
  - Clinical Research & Consulting Center, LLC, Fairfax, Virginia
- Germany (8):
  - KfH Nierenzentrum/Bad/Konig, Bad König
  - KfH Nierenzentrum, Berlin
  - KfH Dialysezentrum/Berlin, Berlin
  - KfH Nierenzentrum/Dulmen, Dülmen
  - Georg-August-Universitat Universitatsmedizin Abt. Nephrologie u. Rheumatologie, Göttingen
  - Dialysezentrum Barmbeck, Hamburg
  - KfH-Nierenzentrum/Jena, Jena
  - KfH-Dialysezentrum/Rosenheim, Rosenheim
- Jose Cangiano, MD, San Juan, Puerto Rico
- Churchill Hospital Oxford Kidney Unit, Oxford, United Kingdom

REFERENCES:
- [Background] Sprague SM, Ross EA, Nath SD, Zhang P, Pratt RD, Krause R. Lanthanum carbonate vs. sevelamer hydrochloride for the reduction of serum phosphorus in hemodialysis patients: a crossover study. Clin Nephrol. 2009 Oct;72(4):252-8. doi: 10.5414/cnp72252. PMID 19825330
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following Washout 1, eligible subjects with serum phosphorus levels greater than or equal to 6.0mg/dL (greater than or equal to 1.94mmol/L) and calcium levels greater than or equal to 8.4mg/dL (greater than or equal to 2.10mmol/L) were randomized in a 1:1 ratio to receive either Fosrenol or sevelamer hydrochloride (HCl) for 4 weeks.
Pre-assignment Details: The study consisted of the following phases: screening (1 week), washout 1 (2 weeks), treatment (4 weeks), Washout 2 (2 weeks), crossover treatment (4 weeks), and a 30-day follow-up
Groups:
- Fosrenol First: Fosrenol (Lanthanum carbonate) dosing began at 2250mg/day, administered orally as one 750mg tablet taken three times per day with meals for 1 week. After receiving this dose for 1 week, subjects received the final dose of 3000mg/day, administered orally as one 1000mg tablet three times per day with meals. Subjects were to remain on the final Fosrenol dose of 3000mg/day for 3 weeks. After washout, patients then crossover to receive Sevelamer HCl for 4 weeks (see below).
- Sevelamer HCl First: Sevelamer HCl dosing began at 4800mg/day, administered orally as two 800mg tablets taken three times per day with meals for 1 week. After receiving this dose for 1 week, subjects received the final dose of 6400mg/day, administered orally as three 800mg tablets taken two times per day with meals and two 800mg tablets taken once per day with the lighter meal (i.e., a total of eight 800mg tablets per day). Subjects were to remain on the final sevelamer HCl dose of 6400mg/day for 3 weeks. After washout, patients then crossover to receive Fosrenol for 4 weeks (see above).
Period: First Intervention
Arm/Group | Fosrenol First | Sevelamer HCl First
Started | 95 | 87
Completed | 77 | 75
Not Completed | 18 | 12
Not completed — Adverse Event | 6 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Kidney transplant | 1 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Subject exceeded safety criteria | 0 | 1
Not completed — Subject met an exclusionary criteria | 1 | 0
Not completed — Extended hospitalization | 1 | 0
Not completed — Site error | 1 | 0
Not completed — Sponsor's request | 1 | 0
Period: Washout
Arm/Group | Fosrenol First | Sevelamer HCl First
Started | 77 | 75
Completed | 77 | 75
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Fosrenol First | Sevelamer HCl First
Started | 77 | 75
Completed | 65 | 68
Not Completed | 12 | 7
Not completed — Adverse Event | 5 | 2
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Kidney Transplant | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Subject exceeded safety criteria | 1 | 0
Not completed — Subject moved | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 140
  >=65 years | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 102
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139
  Puerto Rico | 1
  Germany | 41
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Phosphorus Levels at 4 Weeks
Time Frame: 4 weeks
Population: ITT population defined as subjects who were randomized, received at least one dose of investigational product, and had at least one post-dose assessment of the primary efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Fosrenol: Lanthanum carbonate
Arm/Group | Fosrenol | Sevelamer HCl
Number analyzed (Participants) | 165 | 161
mg/dL | -1.73 (0.129) | -1.44 (0.132)
Statistical Analysis 1: Comparison: Fosrenol vs Sevelamer HCl; Test type: Superiority or Other; p = 0.1130, ANCOVA

2. Secondary Outcome: Change From Baseline in Serum Calcium Levels at 4 Weeks
Time Frame: 4 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Fosrenol | Sevelamer HCl
Number analyzed (Participants) | 165 | 161
mg/dL | 0.06 (0.045) | -0.06 (0.046)
Statistical Analysis 1: Comparison: Fosrenol vs Sevelamer HCl; Test type: Superiority or Other; p = 0.0249, ANCOVA

3. Secondary Outcome: Levels of Intact Parathyroid Hormone (iPTH) at Baseline and 4 Weeks
Time Frame: Baseline and 4 weeks
Population: ITT
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Fosrenol | Sevelamer HCl
Number analyzed (Participants) | 165 | 161
pg/mL
  Baseline | 225.46 (11.094) | 225.46 (11.094)
  Endpoint | 296.48 (17.412) | 291.18 (16.181)

4. Secondary Outcome: Patients Achieving Kidney Disease Outcomes Quality Initiative (KDOQI) Target for Serum Phosphorous at 4 Weeks
Description: Kidney Disease Outcomes Quality Initiative (KDOQI) target for serum phosphorous is 3.5 - 5.5 mg/dL (1.13 - 1.77 mmol/L)
Time Frame: 4 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosrenol | Sevelamer HCl
Number analyzed (Participants) | 165 | 161
Percentage of Participants | 42.7 | 34.6

ADVERSE EVENTS:
Groups:
- Fosrenol: Fosrenol (Lanthanum carbonate) dosing began at 2250mg/day, administered orally as one 750mg tablet taken three times per day with meals for 1 week. After receiving this dose for 1 week, subjects received the final dose of 3000mg/day, administered orally as one 1000mg tablet three times per day with meals. Subjects were to remain on the final Fosrenol dose of 3000mg/day for 3 weeks. After washout, patients then crossover to receive Sevelamer HCl for 4 weeks (see below).
- Sevelamer HCl: Sevelamer HCl dosing began at 4800mg/day, administered orally as two 800mg tablets taken three times per day with meals for 1 week. After receiving this dose for 1 week, subjects received the final dose of 6400mg/day, administered orally as three 800mg tablets taken two times per day with meals and two 800mg tablets taken once per day with the lighter meal (i.e., a total of eight 800mg tablets per day). Subjects were to remain on the final sevelamer HCl dose of 6400mg/day for 3 weeks. After washout, patients then crossover to receive Fosrenol for 4 weeks (see above).
Arm/Group | Fosrenol | Sevelamer HCl
Serious Adverse Events (participants affected / at risk) | 18/170 | 20/163
Other Adverse Events (participants affected / at risk) | 31/170 | 27/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fosrenol (N=170) | Sevelamer HCl (N=163)
Death (Vascular disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1
Foot infection (Infections and infestations) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1
Weakness (General disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Coronary atery disease (Cardiac disorders) | 2 | 2
Osteomyelitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 3 | 1
Extremity necrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Cystitis (Infections and infestations) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Septic phlebitis (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Unstable angina (Cardiac disorders) | 1 | 0
Cerebral vascular accident (Nervous system disorders) | 3 | 0
Pripheral neuropathy (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fosrenol (N=170) | Sevelamer HCl (N=163)
Nausea (Gastrointestinal disorders) | 15 | 9
Diarrhea (Gastrointestinal disorders) | 12 | 12
Vomiting (Gastrointestinal disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.